CLINICAL TRIAL: NCT00197301
Title: Phase 1 Study to Examine the Safety and Efficacy of a Novel Liposomal Based Intranasal Influenza Vaccine
Brief Title: Liposomal Based Intranasal Influenza Vaccine:Safety and Efficacy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-05.08.05-HMO-CTIL
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2005-09

CONDITIONS: Influenza
Keywords: Intranasal vaccination, Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Vaccination

INTERVENTIONS:
Biological: Vaccination

SUMMARY:
Influnza vaccination is highly recommended over the age of 50,but is only 50% efficatious among the elderly. A Vaccine given as a nasal spray may improve compliance and local immunity.Liposomes are lipid particles that may serve as carriers for the vaccine and together they enhance the local immune response in mice when given as nasal spray.This study aims to examine the safety and nasal and humoral responses to the nasal vaccine compared to the commercial muscular vaccine.

ELIGIBILITY:
Inclusion Criteria:Healthy young(20-45years old) and elderly(65-95 years old) volunteers -

Exclusion Criteria:Known allergy to eggs and to the flu vaccine, pregnant and breast feeding women, chronic viral carriers, recently hospitalized persons

-

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-10; Study Completion 2006-04

PRIMARY OUTCOMES:
Seroprotection

SECONDARY OUTCOMES:
Antibody levels

CONTACTS AND LOCATIONS:
Overall Officials: Arie Ben Yehuda, M.D., Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel